CLINICAL TRIAL: NCT01661374
Title: The Effect of Humidification on Mucus Rheology
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: HM14433
Record Dates: First submitted 2012-08-06; First posted 2012-08-09 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease(COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mechanically Ventilated
- Chronic obstructive pulmonary disease (COPD).

SUMMARY:
In this study the investigators will collect mucus from mechanical ventilated patients and patients with COPD to study the effect of temperature and humidity, on the biophysical properties of the airway mucus. It is hypothesised that changes in inspired gas temperature and humidity (over time) may affect the biophysical properties of the airway mucus and reduce the airway's ability to clear mucus, resulting in deleterious clinical affects.

DETAILED DESCRIPTION:
Expectorated sputum samples are collected and used to measure the biophysical properties of mucus secretions. The samples are later exposed to different temperatures and humidity levels during bench experiments.

ELIGIBILITY:
Mechanically Ventilated Patients

Inclusion Criteria:

Any Subject Mechanically Ventilated and producing sputum.

Exclusion

* None

COPD Group

Inclusion Criteria:

* 40 to 90 years of age suffering from COPD
* History of mucus production

Exclusion Criteria:

* None

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic,ICU, Pulmonary Clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sputum Collection | 10 minutes
  Sputum is collected during pulmonary function test (PFT) to later measure the biophysical properties of sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MEngr, MD, MBA, FRCPC, Principal Investigator — Virginia Commonwealth University School of Medicine
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States